CLINICAL TRIAL: NCT05556681
Title: Prospective, Multicenter, Single Arm, Non-Randomized Study of BD Sirolimus Drug Coated Catheter for Treatment of Femoropopliteal Arteries
Brief Title: Study of BD Sirolimus Drug Coated Catheter for Treatment of Femoropopliteal Arteries
Acronym: PREVISION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BDPI-20-012
Record Dates: First submitted 2022-09-12; First posted 2022-09-27 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Peripheral Arterial Disease; Peripheral Artery Disease; Stenosis Artery
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treated with the investigational BD™ Sirolimus Drug Coated Catheter (Experimental): Patients treated with the BD™ Sirolimus Drug Coated Catheter
  Interventions: Device: BD™ Sirolimus Drug Coated Balloon Catheter percutaneous transluminal angioplasty

INTERVENTIONS:
Device: BD™ Sirolimus Drug Coated Balloon Catheter percutaneous transluminal angioplasty — The study will enroll patients presenting with clinical evidence of an angiographically significant lesion (Lesion ≥ 70% stenosis by visual estimate) in the femoropopliteal arteries. Eligible patients will undergo percutaneous transluminal angioplasty with the investigational BD™ Sirolimus Drug Coated Balloon Catheter.

SUMMARY:
The objective of this early feasibility study is to assess the safety and performance of the BD™ Sirolimus Drug Coated Balloon Catheter.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized, single-arm early feasibility study designed to assess the safety and performance of the BD™ Sirolimus Drug Coated Balloon Catheter for the treatment of stenosis in the femoropopliteal arteries. Follow-up for all treated subjects will be performed at post-procedure, 30 days, and 6, 12 months, 18 months and 24 months post-index procedure.

ELIGIBILITY:
Inclusion Criteria:

Pre-Operative Inclusion Criteria:

1. ≥18 years of age.
2. Rutherford Clinical Category 2-4.
3. Participant is willing to provide informed consent, is geographically stable, comply with the required follow up visits and testing schedule and recommended medication regimen.
4. Women of childbearing potential who have a negative UPT at screening.

   Angiographical Inclusion Criteria:
5. One Lesion of ≥ 3 cm and ≤ 17 cm in length (if two discrete lesions are separated by ≤ 3 cm, but both falling within a composite length of ≤ 17 cm, they may be treated as one lesion).
6. Lesion ≥70% stenosis by visual estimate.
7. Lesion location starts ≥1 cm below the common femoral bifurcation and terminates above the distal P2 segment (top of the tibial plateau).
8. De novo or non-stented restenotic lesion(s) in native femoropopliteal arteries >90 days from prior interventional procedure.
9. Lesion is located at least 3 cm from any stent.
10. Target reference vessel diameter of 5-6 mm and able to be treated with available device size matrix.
11. Successful, uncomplicated (without use of crossing device, specialty 035 guidewires are acceptable) antegrade wire crossing of lesion.
12. Successful vessel preparation of the target lesion. Successful vessel preparation is defined by successful pre-dilatation to nominal of the target lesion, in the absence of early recoil, significant residual stenosis ≤30% as confirmed by angiography without any major vascular complications or flow-limiting dissections.
13. A patent inflow artery free from significant lesion stenosis (≥50% stenosis) as confirmed by standard of care imaging and the discretion of the investigator Only treatment of ipsilateral iliac inflow arteries is acceptable before the treatment of the target lesion, defined as attainment of residual diameter stenosis ≤30% without death or major vascular complication.
14. At least one patent native outflow artery to the ankle, free from significant (≥50%) stenosis as confirmed by angiography, that has not previously been revascularized (outflow to be assessed after successful vessel preparation of target lesion; treatment of outflow disease is NOT permitted during the index procedure).

Exclusion Criteria:

Pre-Operative Exclusion Criteria:

1. ≥ 90 years of age.
2. Women who are breastfeeding, currently pregnant or planning to become pregnant during the duration of the study or have a positive urine pregnancy test at screening. Men who are intending to biologically father children during the duration of the study.
3. Life expectancy of <2 years
4. Participant has acute limb ischemia.
5. Previous treatment of the target limb using Drug Coated Balloon (DCB), a stent, or Drug Eluting Stent (DES) within the last 180 days.
6. Previous treatment of the contralateral limb using Drug Coated Balloon (DCB) or Drug Eluting Stent (DES) within the last 90 days.
7. History of stroke or TIA within 90 days.
8. History of myocardial infarction (MI), thrombolysis or angina within 30 days of index procedure.
9. Renal failure (on dialysis) or chronic kidney disease (Glomerular Filtration Rate (GFR) < 30 ml/min per 1.73m2 (or serum creatinine ≥2.5 mg/L within 30 days of index procedure or treated with dialysis)) that in the opinion of the investigator should preclude participant enrollment in the study.
10. Active or suspected active infection at time of index procedure that in the opinion of the investigator should preclude participant enrollment in the study.
11. Patients with any type of previous or planned surgical or interventional procedure within 30 days prior and/or within 30 days post-index procedure.
12. Sudden symptom onset (within two weeks), acute vessel occlusion, or acute or sub-acute thrombus in target vessel or history of treatment of thrombolysis in the target lesion.
13. Known contraindication (including allergic reaction) or sensitivity to sirolimus (rapamycin).
14. Known contraindication (including reaction) or sensitivity to iodinated contrast media, that cannot be adequately managed with pre- and post-procedure medication. CO2 angiography is not allowed.
15. Has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 3 months prior to Screening (for corticosteroids ≥ 20 mg/day of prednisone equivalent, excluding standard of care use of inhaled corticosteroids).
16. Immunosuppressive or immunodeficient state, in the opinion of the investigator, that would preclude the participant from being eligible to be treated with a sirolimus DCB. Note: HIV positive participants with CD4 count ≥350 cells/mm3 and an undetectable HIV viral load within the past year [low level variations from 50-500 viral copies which do not lead to changes in antiretroviral therapy [ART] are permitted.
17. Has active malignancy prior to study entry.
18. Bleeding diathesis, Gastrointestinal ulceration, another coagulopathy disorder, or allergy in the opinion of the investigator, which would restrict the use of anticoagulant or dual antiplatelet therapy (DAPT).
19. Participant is currently participating in an investigational drug or device study, or previously enrolled in this study. Enrollment in another investigational drug or device study during the follow up period for this study is not allowed.
20. Current alcohol or drug abuse that in the opinion of the investigator should preclude participant enrollment in the study.
21. Participant has a condition that in the opinion of the investigator should preclude participant enrollment in the study.

    Angiographical Exclusion Criteria:
22. Severe Calcification as defined as PARC scoring system (> 180 degrees (both sides of the vessel at the same location) and greater than one-half of the total lesion length) of the target lesion.
23. Intended use of adjunctive primary treatment modalities (e.g., atherectomy, laser, cutting balloons, radiation therapy, stents, other drug coated devices.)
24. Use of reentry devices during the index procedure for antegrade recanalization, which include but are not limited to percutaneous intentional extraluminal recanalization (PIER) and subintimal arterial flossing with antegrade retrograde intervention (SAFARI) techniques.

Pharmacokinetic (PK) Sub-Study:

Inclusion Criteria:

1. Participant must meet all main study inclusion and exclusion criteria.

Exclusion Criteria:

1. Previous treatment or planned treatment with any Drug Coated Balloon (DCB) or Drug Eluting Stent (DES) in the last 12 months and within 6 months post study index procedure.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Late lumen loss at six months as measured by quantitative vascular angiography (QVA). | at 6 month follow-up
  Late lumen loss is defined as the difference (in mm) between the minimum lumen diameter (MLD) of the treated segment at follow up and the measurement immediately after the index procedure.

SECONDARY OUTCOMES:
Rutherford Improvement | at discharge, and 1, 6, 12 and 24 month follow-up
  This endpoint will be evaluated by descriptive statistics and will not have statistical analyses associated with them but will be reported upon in the final study report.
Patient Reported Outcome Improvement | at post-procedure, and 1, 6, 12 and 24 month follow-up
  This endpoint will be evaluated by descriptive statistics and will not have statistical analyses associated with them but will be reported upon in the final study report.
Freedom of Embolization | at discharge, and 1, 6, 12 and 24 month follow-up
  This endpoint will be evaluated by descriptive statistics and will not have statistical analyses associated with them but will be reported upon in the final study report.
ABI Improvement | at discharge, and 1, 6, 12 and 24 month follow-up
  This endpoint will be evaluated by descriptive statistics and will not have statistical analyses associated with them but will be reported upon in the final study report.
Revascularization rate (CD-TLR) | at discharge, and 1, 6, 12 and 24 month follow-up
  This endpoint will be evaluated by descriptive statistics and will not have statistical analyses associated with them but will be reported upon in the final study report.
Technical & Procedural Success statistical analyses associated with them but will be reported upon in the final study report. | at discharge, and 1, 6, 12 and 24 month follow-up
  This endpoint will be evaluated by descriptive statistics and will not have statistical analyses associated with them but will be reported upon in the final study report.
All Cause Death statistical analyses associated with them but will be reported upon in the final study report. | at discharge, and 1, 6, 12 and 24 month follow-up
  This endpoint will be evaluated by descriptive statistics and will not have statistical analyses associated with them but will be reported upon in the final study report.
Major Adverse Cardiovascular Events (MACE) statistical analyses associated with them but will be reported upon in the final study report. | at discharge, and 1, 6, 12 and 24 month follow-up
  This endpoint will be evaluated by descriptive statistics and will not have statistical analyses associated with them but will be reported upon in the final study report.
Safety Composite statistical analyses associated with them but will be reported upon in the final study report. | at discharge, and 1, 6, 12 and 24 month follow-up
  This endpoint will be evaluated by descriptive statistics and will not have statistical analyses associated with them but will be reported upon in the final study report.

CONTACTS AND LOCATIONS:
Overall Officials: Talar Saber, Study Director — Becton, Dickinson and Company (BD) (CRBARD)
Locations (10):
- Australia (6):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - Flinders University, Adelaide, South Australia
  - The Alfred, Melbourne, Victoria
  - Royal Perth Hospital, Perth, Western Australia
- New Zealand (2):
  - Auckland City Hospital, Grafton, Auckland
  - Waikato Hospital, Hamilton, Waikato Region
- Singapore (2):
  - Tan Tock Seng Hospital, Novena
  - Sengkang General Hospital, Punggol

IPD SHARING:
Plan to Share IPD: No
Data in aggregate